CLINICAL TRIAL: NCT07298590
Title: An Exploratory Clinical Study on the Safety and Efficacy of CD19/BCMA CAR-NK (KN5601) in the Treatment of Relapsed and Refractory IgG4-related Disease (IgG4-RD)
Brief Title: An Exploratory Clinical Study on the Safety and Efficacy of CD19/BCMA CAR-NK in the Treatment of Relapsed and Refractory IgG4-related Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2025-364; CHEC2025-473 (Other: Shanghai Changhai Hospital)
Record Dates: First submitted 2025-11-17; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: IgG4 Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This study is a single-arm, open-label and single-center exploratory clinical study (Experimental)
  Interventions: Biological: CD19/BCMA CAR NK

INTERVENTIONS:
Biological: CD19/BCMA CAR NK — Patients will receive Fludarabine and Cyclophosphamide on day -5, -4, and -3. Multiple doses of CD19/BCMA CAR NK cells will infused using the dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of CD19/BCMA CAR NK cells (KN5601) in patients with IgG4 related diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and provide informed consent and be willing to comply with study procedures and follow-up.
2. The age at the time of signing the informed consent must be at least 18 years old and no more than 70 years old.
3. Meet the 2020 Japanese criteria or ACR/EULAR IgG4-RD classification criteria.
4. Subjects with relapsed/refractory active IgG4-RD at screening on an IgG4-RD RI ≥4, simultaneously meeting the following definitions of relapse or refractory disease:

   1. Definitions of relapse: subjects with IgG4-RD achieved remission after treatment but was active again before screening, and were classified as a high-risk group for recurrence assessed by assessment committee ;
   2. Definitions of before screening: subjects had used glucocorticoids or glucocorticoids combined with at least one conventional synthetic disease-modifying antirheumatic drug (csDMARDs) (including cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide, elorimod, thalidomide, etc.), or at least one approved biologic agent (bDMARDs) (including rituximab, abatacept, etanercept, belimumab, etc.), or targeted synthetic (ts) DMARDs (including tofacitinib, upadacitinib, baricitinib, abrocitinib, deucravacitinib, etc.) for treatment, with a total treatment duration of ≥3 months, yet still in an active disease state, ineffective, intolerant, or experiencing relapse during glucocorticoid tapering.
5. No history of severe allergic reaction.
6. Female participants of childbearing age must have a negative pregnancy test upon enrollment in the study; indeterminate results will not be accepted.
7. Female subjects of childbearing age and male subjects with female partners of childbearing potential must agree to consistently use effective methods of birth control within 6 months after the last KN5601 infusion.
8. Echocardiography show that the heart structure is basically normal and the left ventricular ejection fraction (LVEF) is ≥55%; no obvious abnormalities are found on the electrocardiogram.
9. Pulmonary function: No severe lung disease, SpO2 ≥ 92%.
10. All subjects' eligibility for enrollment must be confirmed by an independent Assessment Committee (AC) (the committee consists of independent data monitors and clinical experts separate from the study). They will review the eligibility of each patient based on the scores entered at screening, as well as brief descriptions provided by the investigators regarding the supporting diagnosis, scores, and the patient's clinical status in relation to enrollment criteria..

Exclusion Criteria:

1. Presence of a condition other than IgG4-RD that (e.g., asthma) is likely to require systemic Glucocorticoids (GC) for disease control during the period of the trial.
2. Malignancy within 5 years (except successfully treated in situ cancer, resected squamous cell or basal cell carcinoma of the skin.).
3. During the screening visit, one of the following laboratory test values must be met, except for those caused by IgG4-RD.:

   1. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than three times the upper limit of normal (ULN).
   2. Total bilirubin > two times the ULN unless caused by Gilbert's disease. Gilbert's disease with total bilirubin > three times ULN.
   3. White blood cell (WBC) count <3.0×10⁹/L;
   4. Absolute neutrophil count (ANC) <1.5×10⁹/L;
   5. Hemoglobin <90 g/L;
   6. Platelet count <75×10⁹/L;
   7. Estimated glomerular filtration rate (eGFR) ≤ 45 ml/(min·1.73m2).
4. Evidence suggests the presence of another uncontrolled disease, which the investigator has determined may affect the subject's participation in the trial.
5. Active infection requiring hospitalization or treatment with systemic antimicrobial agents within the 30 days prior to treatment allocation/randomization.
6. Received rituximab or other B-cell depleting therapies within 6 months prior to the baseline visit, unless B cells have recovered (B-cell recovery is defined as peripheral blood B-cell count ≥ the lower limit of normal reference range or returned to pre-treatment levels)。
7. The use of supplemental oxygen at baseline.
8. During the screening visit or within 90 days prior to the screening visit: T-SPOT positive. If the result is indeterminate, the T-SPOT must be repeated (using the same or a different T-SPOT) and shown as negative.
9. During screening visits, individuals with a history of chronic infection or serological evidence, including:

   1. Human immunodeficiency virus infection;
   2. Hepatitis B as indicated by surface antigen or hepatitis B core antibody positivity;
   3. Hepatitis C as indicated by anti-hepatitis C antibody positivity; if a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if he/she is negative for viral load at screening.
10. Planned vaccination with live vaccines during the trial.
11. Participant is pregnant or breastfeeding, or planning a pregnancy while enrolled in the study.
12. IgG4-RD that is dominated primarily by advanced fibrotic lesions. Specifically, participants whose disease manifestations consist only of

    1. retroperitoneal fibrosis,
    2. fibrosing mediatinitis,
    3. sclerosing mesenteritis, and
    4. Riedel's thyroiditis. Subjects were eligible to be included only if they had non-advanced fibrotic disease in at least one organ system and otherwise met the inclusion and exclusion criteria.
13. Evidence a SARS-CoV-2 (COVID-19) infection started within the 30 days prior to treatment allocation/randomization. Participants diagnosed with SARS-CoV-2 (COVID-19) infection more than 30 days prior to treatment .allocation/randomization must have symptoms resolved and be deemed fit to participate in the trial.
14. Researchers consider any situations that may increase the risk to participants or interfere with the trial results (including but not limited to a history of mental illness, alcoholism, drug abuse, poor compliance, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06-26 (Estimated); Study Completion 2028-12-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 48 weeks
  To characterize the safety of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 48 weeks
  To characterize the safety of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
The percentage of disease remission (Remission is defined as IgG4-RD RI=0 after treatment and without the use of hormones | 24 weeks
  To characterize the safety of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases

SECONDARY OUTCOMES:
Percentage of disease remission of IgG4-RD RI score compared with baseline | 12, 24, 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Percentage of complete response, partial response, and no change (NC) | 12, 24, 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Disease recurrence rate | 24, 48 weeks after infusion
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Physician Global Assessment (PhGA) compared with baseline | up to 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related disease
Patient Global Assessment (PGA) compared with baseline | 12, 24, 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related disease
Disease-related Injury Score | 12, 24, 48 weeks
  To characterize the safety of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Health Survey by Health Status Questionnaire (SF-36) | up to 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Assessment of organ function compared with baseline based on MRl imaging | up to 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Assessment of the affected tissues and organs compared with baseline based on CT imaging examination | up to 48 weeks
  To characterize the efficacy of CD19/BCMA CAR NK Cells (KN5601) for IgG4 related diseases
Assessment of persistence of KN5601 after infusion | up to 48 weeks
  To detect CAR copy numbers of KN5601 in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No